CLINICAL TRIAL: NCT00799448
Title: Multi-centre, Open, Randomised, Parallel, Controlled Trial in Type 2 Diabetic Subjects Inadequately Controlled With SU +/ Biguanide Therapy, to Compare the Efficacy and Safety of Repaglinide Combined With Bedtime Insulin vs. Insulin Alone
Brief Title: Comparison of Efficacy and Safety of Repaglinide Combined With Insulin NPH Versus Biphasic Human Insulin 30 Alone in Inadequately Controlled Subjects With Type 2 Diabetes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment status
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGEE-1524
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; biphasic human insulin 30; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: repaglinide
Drug: biphasic human insulin 30
Drug: insulin NPH

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the efficacy and safety of repaglinide combined with insulin NPH versus biphasic human insulin 30 alone in type 2 diabetics inadequately controlled with sulfonylurea (SU) +/ biguanide therapy

ELIGIBILITY:
Inclusion Criteria:

* HbA1c: 7.5-11.0% on current therapy
* OHA (oral hypoglycaemic agent) treatment for a minimum of two years
* BMI (body mass index): 25-32 kg/m2

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-09-16 (Actual); Primary Completion 2004-09-20 (Actual); Study Completion 2004-09-20 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 20 weeks of treatment

SECONDARY OUTCOMES:
Fasting blood glucose (FBG)
Incidence of hypoglycaemic episodes
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Athens, Greece

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com